CLINICAL TRIAL: NCT02574533
Title: A Pilot Study of Vigil™ Augmented Autologous Tumor Cell Immunotherapy in Combination With Pembrolizumab PD-1 Inhibitor for Patients With Advanced Melanoma
Brief Title: Pilot Study of Vigil™ + Pembrolizumab for Advanced Melanoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Gradalis, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CL-PTL-123
Record Dates: First submitted 2015-10-09; First posted 2015-10-14 (Estimated); Last update posted 2017-09-27 (Actual); Status verified 2017-09

CONDITIONS: Melanoma Recurrent; Malignant Melanoma; Melanoma
Keywords: Immunotherapy; PD-1 inhibitor; Keytruda; checkpoint inhibitor; vaccine; FANG; Vigil
MeSH Terms: conditions — Melanoma | interventions — FANG vaccine; pembrolizumab; Immune Checkpoint Inhibitors

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Vigil™ + Pembrolizumab (Experimental): Biological: Vigil™ 1 x 10e7 cells via intradermal injection on Day 1, 15, 29, 43 and then every 3 weeks thereafter for a minimum of 4 administrations and a maximum of 9 administrations (depending on the quantity of Vigil™ manufactured from surgical specimens.
  Drug: Pembrolizumab 2mg/kg by intravenous infusion over 30 minute starting on day 43 and every 3 weeks thereafter
  Interventions: Biological: Vigil; Drug: Pembrolizumab

INTERVENTIONS:
Biological: Vigil — Vigil™ 1 x 10e7 cells via intradermal injection on Day 1, 15, 29, 43 and then every 3 weeks thereafter for a minimum of 4 administrations and a maximum of 9 administrations (depending on the quantity of Vigil™ manufactured from surgical specimens)
  Other Names: formerly known as FANG™; bi-shRNAfurin and GMCSF Autologous Tumor Cell Immunotherapy
Drug: Pembrolizumab — Pembrolizumab 2mg/kg by intravenous infusion over 30 minute starting on day 43 and every 3 weeks thereafter
  Other Names: Keytruda®; PD-1 inhibitor

SUMMARY:
This is an open label Pilot study to evaluate the combination of Vigil™ and pembrolizumab in patients with incurable locally advanced or metastatic melanoma. Patients undergoing a standard of care surgical procedure (e.g., tumor biopsy, palliative resection) and meeting procurement eligibility criteria may have tumor harvested for Vigil™ vaccine manufacture. This study evaluates the hypothesis that vaccination with Vigil™ will induce cancer-specific T cell immunity in these patients. Addition of pembrolizumab to Vigil™ treated patients will further augment these immune changes on sequential biopsy when comparing post-Vigil™ but pre-PD-1 inhibitor to post-PD-1 inhibitor biopsies, and the combination therapy will be associated with reduction of tumor volume on clinical exam and/or imaging.

DETAILED DESCRIPTION:
This is an open label Pilot study to evaluate the combination of Vigil™ autologous tumor cell immunotherapy and pembrolizumab PD-1 inhibitor in patients with incurable locally advanced or metastatic melanoma. Patients undergoing a standard of care surgical procedure (e.g., tumor biopsy, palliative resection) and meeting procurement eligibility criteria may have tumor harvested for Vigil™ vaccine manufacture. Patients subsequently meeting study enrollment criteria including manufacture of a minimum of 4 doses of Vigil™ and agreement to provide on treatment tumor biopsies will receive (i) Vigil™ 1 x 10e7 cells intradermal on Days 1, 15, 29, 43 and every 3 weeks thereafter for up to 9 total doses of Vigil™ and (ii) pembrolizumab 2 mg/kg IV starting on Day 43 and every 3 weeks thereafter for up to 6 months from study enrollment. Day 1 of study treatment must be within 6 weeks of tumor procurement. Tumor biopsy and peripheral blood mononuclear cells (PBMCs) for correlative studies will be obtained at baseline (before tumor procurement), and at Week 7 and Week 16 while on study. PBMCs will also be collected at Week 1 (pre-Vigil™) and end of treatment (EOT). Radiological assessment of tumor by immune related Response Criteria (irRC) and RECIST criteria will be obtained at screening (after tumor procurement) and at Week 13 and EOT.

The primary study objective is to characterize and compare CD8+ T cell density, PD-1+ T cell density, and PD-L1 expression on tumor biopsy at baseline, following 3 doses (approximately 6 weeks) of single agent Vigil™ and again following 3 doses of pembrolizumab. Secondary study objectives include evaluation of tolerability and safety of the combination, and to determine and compare IFNγ-ELISPOT result pre-procurement, at screening, after single agent Vigil™, and after Vigil™ plus pembrolizumab combination. Additional study objectives include determining best ORR by irRC criteria.

ELIGIBILITY:
Tissue Procurement Inclusion Criteria:

Patients will be eligible for tissue procurement for the Vigil™ manufacturing process, if they meet all of the following criteria:

1. Age ≥ 18 years.
2. ECOG Performance Status ≤ 1
3. Estimated survival ≥ 6 months.
4. If activating BRAF mutation present, subject has previously received BRAF and/or MEK inhibitor
5. Planned standard of care surgical procedure (e.g., tumor biopsy or palliative resection or thoracentesis) and expected availability of a cumulative mass of ~10-30 grams tissue ("golf-ball" size) for vaccine manufacture. Tissue obtained for vaccine manufacture must not have been previously irradiated.
6. At least one area of cancer that is not intended for resection or vaccine manufacture and in the opinion of the investigator is appropriate for serial biopsy.
7. Ability to understand and the willingness to sign a written informed consent document for tissue harvest.

Tissue Procurement Exclusion Criteria:

Patients meeting any of the following criteria are not eligible for tissue procurement for the Vigil™ manufacturing:

1. Documented history of tumor PD-L1 expression positivity (defined as membranous staining of neoplastic cells >1%)
2. Anti-cancer chemotherapy, immunotherapy, or biologic therapy within 3 weeks or radiation therapy within 1 week prior to procurement of tumor for vaccine manufacture.
3. Radiation therapy treatment of lesion intended for vaccine manufacture unless post-radiation progression of that lesion is confirmed.
4. Medical condition requiring any form of chronic systemic immunosuppressive therapy (steroid or other) except physiologic replacement doses of hydrocortisone or equivalent (no more than 30 mg hydrocortisone or 10 mg prednisone equivalent daily) for < 30 days duration
5. Known history of other malignancy unless having undergone curative intent therapy without evidence of that disease for ≥ 3 years except cutaneous squamous cell and basal cell skin cancer, superficial bladder cancer, in situ cervical cancer or other in situ cancers are allowed if definitively resected.
6. Brain metastases unless treated with curative intent (gamma knife or surgical resection) and without evidence of progression for ≥ 2 months.
7. Any documented history of autoimmune disease with exception of Type 1 diabetes on stable insulin regimen, hypothyroidism on stable dose of replacement thyroid medication, vitiligo, or asthma not requiring systemic steroids.
8. Known history of allergies or sensitivities to gentamicin.
9. History of or current evidence of any condition (including medical, psychiatric or substance abuse disorder), therapy, or laboratory abnormality that might confound the results of the study, interfere with the patient's participation for the full duration of the study, or is not in the best interest of the patient to participate, in the opinion of the treating Investigator.
10. Known HIV or chronic Hepatitis B or C infection.
11. History of pneumonitis or interstitial lung disease.

Study Enrollment Inclusion Criteria:

Patients will be eligible for registration into the trial if they meet all of the following inclusion criteria:

1. Successful manufacturing of at least 4 vials of Vigil™.
2. ECOG performance status (PS) ≤ 1
3. Estimated survival ≥ 4 months.
4. Adequate organ function as defined by the following laboratory values:

   * Hematological Absolute granulocyte count ≥ 1,500/mm3
   * Hematological Absolute lymphocyte count ≥ 500/mm3
   * Hematological Platelets ≥ 75,000/mm3
   * Hematological Hemoglobin ≥ 9 g/dL
   * Renal Creatinine ≤ 1.5x institutional upper limit of normal
   * Hepatic Total bilirubin ≤ 1.5x institutional upper limit of normal
   * Hepatic AST(SGOT) and ALT(SGPT) ≤2x institutional upper limit of normal or

     ≤5x institutional upper limit of normal if liver metastases
   * Coagulation INR / PT and aPTT ≤ 1.5 x ULN (if not using anticoagulants)*If patient receiving anticoagulant therapy value must be within therapeutic range for the condition being treated.
   * Immunological Thyroid Stimulating Hormone within institutional limits**If TSH is greater or less than institutional limits patients may participate if their T4 is within normal limits (WNL); patients may be on a stable dose of replacement thyroid medication; dose adjustments are allowed if needed.
5. Subject has recovered to CTCAE Grade 1 or better from all adverse events associated with prior therapy or surgery. Pre-existing motor or sensory neurologic pathology or symptoms must be recovered to CTCAE Grade > 2 or better.
6. If female of childbearing potential, has a negative urine or serum pregnancy test. If the urine test is positive or cannot be confirmed as negative, a negative serum test will be required for study entry.
7. Patient has agreed to provide on study tumor biopsies for correlative research.
8. Ability to understand and the willingness to sign a written informed protocol specific consent.

Study Enrollment Exclusion Criteria:

In addition to the procurement exclusion criteria, patients will NOT be eligible for study registration and enrollment if meeting any of the following criteria:

1. Any anti-neoplastic therapy between tissue procurement for vaccine manufacture and start of study therapy.
2. Live vaccine used for the prevention of infectious disease administered < 30 days prior to the start of study therapy.
3. Post-surgery complication that in the opinion of the treating investigator would interfere with the patient's study participation or make it not in the best interest of the patient to participate.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2015-10 (Actual); Primary Completion 2017-09 (Actual); Study Completion 2017-09 (Actual)

PRIMARY OUTCOMES:
Tumor Immune-Related Response to Vigil and Vigil + Pembrolizumab | 16 weeks
  Tumor Immune-Related Response to Vigil and Vigil + Pembrolizumab as measured by Tumor biopsy for Immunohistochemistry

SECONDARY OUTCOMES:
Best Overall Response Rate (ORR) to Vigil and Vigil + Pembrolizumab | 26 weeks
  Best Overall Response Rate (ORR) to Vigil and Vigil + Pembrolizumab as measured by:
  * Radiological Tumor Assessment (irRC) and Response Evaluation Criteria in Solid Tumors (RECIST) Version 1.1.
  * IFNγ-ELISPOT conversion rate
Toxicities and AEs for Vigil + Pembrolizumab according to the Common Toxicity Criteria for Adverse Events (CTCAE) Version 4.03 | 26 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Luisa Manning, MD, Study Director — Gradalis, Inc.
Locations (3):
- United States (3):
  - Texas Oncology P.A., Texas Cancer Center, Abilene, Texas
  - Mary Crowley Medical Research Centers, Dallas, Texas
  - Cancer Care Northwest, Spokane, Washington

REFERENCES:
- [Background] Nemunaitis J, Barve M, Orr D, Kuhn J, Magee M, Lamont J, Bedell C, Wallraven G, Pappen BO, Roth A, Horvath S, Nemunaitis D, Kumar P, Maples PB, Senzer N. Summary of bi-shRNA/GM-CSF augmented autologous tumor cell immunotherapy (FANG) in advanced cancer of the liver. Oncology. 2014;87(1):21-9. doi: 10.1159/000360993. Epub 2014 Jun 25. PMID 24968881
- [Background] Senzer N, Barve M, Kuhn J, Melnyk A, Beitsch P, Lazar M, Lifshitz S, Magee M, Oh J, Mill SW, Bedell C, Higgs C, Kumar P, Yu Y, Norvell F, Phalon C, Taquet N, Rao DD, Wang Z, Jay CM, Pappen BO, Wallraven G, Brunicardi FC, Shanahan DM, Maples PB, Nemunaitis J. Phase I trial of "bi-shRNAi(furin)/GMCSF DNA/autologous tumor cell" vaccine (FANG) in advanced cancer. Mol Ther. 2012 Mar;20(3):679-86. doi: 10.1038/mt.2011.269. Epub 2011 Dec 20. PMID 22186789
- [Background] Ghisoli M, Barve M, Mennel R, Lenarsky C, Horvath S, Wallraven G, Pappen BO, Whiting S, Rao D, Senzer N, Nemunaitis J. Three-year Follow up of GMCSF/bi-shRNA(furin) DNA-transfected Autologous Tumor Immunotherapy (Vigil) in Metastatic Advanced Ewing's Sarcoma. Mol Ther. 2016 Aug;24(8):1478-83. doi: 10.1038/mt.2016.86. Epub 2016 Apr 25. PMID 27109631
- [Background] Ghisoli M, Barve M, Schneider R, Mennel R, Lenarsky C, Wallraven G, Pappen BO, LaNoue J, Kumar P, Nemunaitis D, Roth A, Nemunaitis J, Whiting S, Senzer N, Fletcher FA, Nemunaitis J. Pilot Trial of FANG Immunotherapy in Ewing's Sarcoma. Mol Ther. 2015 Jun;23(6):1103-1109. doi: 10.1038/mt.2015.43. Epub 2015 Mar 19. PMID 25917459